CLINICAL TRIAL: NCT02802488
Title: Age Related D-dimer Evaluation for the Exclusion of a Left Atrium Thrombus in Patients With Atrial Fibrillation (ADDIT-AF)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brugmann University Hospital (Other)
Responsible Party: Principal Investigator, José Castro, Head of clinic, Brugmann University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHUB-ADDIT-AF
Record Dates: First submitted 2016-06-13; First posted 2016-06-16 (Estimated); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Atrial Fibrillation
Keywords: D-dimers; Atrial fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- D-dimers (Experimental): This arm encompasses patients between 18 and 80 years old and diagnosed with atrial fibrillation.
  Interventions: Procedure: Blood sampling

INTERVENTIONS:
Procedure: Blood sampling — A blood sampling will be performed in patients diagnosed with atrial fibrillation in order to test if having a D-dimers value superior or equal to the patient's age is predictive of a thrombus.
  Thombus will be diagnosed according to the standard of care.

SUMMARY:
Patients with atrial fibrillation are at increased risk of thrombus formation in the left heart, especially in the auricula and the atrium. Their presence increases the risk of ischemic stroke, especially during cardioversion, performed either by drug or by external electric shock. The gold standard to exclude this thrombus and consider cardioversion is the transesophageal echocardiography.

D-dimers, products of the degradation of fibrin, have been studied several times to assess the presence of thrombi in the body, especially in pulmonary embolism. In cardiology and despite several studies on the matter, there is currently no blood D-dimers value allowing to detect the presence of a thrombus with a good predictive value. Correlating the D-dimer values with age, as has been done for some years in pulmonary embolism, would give the opportunity to create a simple, inexpensive and widely applicable tool to eliminate the presence of a thrombus in the left heart.

If the results are satisfactory, the investigators might consider not using transesophageal echocardiography as this examination is unpleasant for the patient and operator dependant, unlike a standard blood sampling.

This study aims to test the following hypothesis: D-dimers values superior or equal to ten times the patient's age is predictive of a thrombus.

ELIGIBILITY:
Inclusion Criteria:

* Patients with de novo or recent atrial fibrillation requiring cardioversion, either by drug, by an electric shock or an intervention.

Exclusion Criteria:

* valvulopathy
* infection
* neoplasia
* inflammatory disease
* recent surgery
* pregnancy
* aorta aneurism
* deep vein thrombosis
* pulmonary embolism

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2020-05-14 (Actual); Study Completion 2020-05-14 (Actual)

PRIMARY OUTCOMES:
D-dimers concentration | first day of hospitalization
  Concentration of D-dimers in the blood

CONTACTS AND LOCATIONS:
Overall Officials: José Castro, MD, Principal Investigator — CHU Brugmann; Alexandre Almorad, MD, Principal Investigator — CHU Brugmann
Locations (1):
- CHU Brugmann, Brussels, Belgium